CLINICAL TRIAL: NCT02528019
Title: Effects of the DPP-4 or SGLT2 Inhibitors on the Metabolic Cardiovascular Systems in Patients With Type 2 Diabetes Mellitus.
Brief Title: Metabolic and Cardiovascular Effects of Dipeptidyl Peptidase-4 (DPP-4) or Sodium-glucose Co-transporter Type 2 (SGLT2) Inhibitors
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kurume University (Other)
Responsible Party: Principal Investigator, Nobuhiro Tahara, Associate Professor, Kurume University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Anti-athero
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Effects of the DPP-4 Inhibitors or SGLT2 Inhibitors on the Protective Actions for Diabetic Complications
MeSH Terms: interventions — Sodium-Glucose Transporter 2 Inhibitors; glimepiride

ARMS (3):
- DPP-4 inhibitors (Active Comparator): sitagliptin (25-100mg daily), vildagliptin (50-100mg daily), alogliptin (12.5-25mg daily), linagliptin (2.5-5mg daily), teneligliptin (20-40mg), anagliptin (100-200mg daily), saxagliptin (2.5-5mg daily) or trelagliptin (50-100mg weekly)
  Interventions: Drug: DPP-4 inhibiotors
- SGLT2 inhibitors (Active Comparator): ipragliflozin (50-100mg daily), dapagliflozin (5-10mg daily), luseogliflozin (2.5-5mg), tofogliflozin (20mg daily), canagliflozin (100mg daily) or empagliflozin (10-25mg daily)
  Interventions: Drug: SGLT2 inhibitors
- Glimepiride (Active Comparator): glimepiride (0.5-8mg daily)
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: DPP-4 inhibiotors
  Arms: DPP-4 inhibitors
Drug: SGLT2 inhibitors
  Arms: SGLT2 inhibitors
Drug: Glimepiride
  Arms: Glimepiride

SUMMARY:
Inhibition of dipeptidyl peptidase-4 (DPP-4) or sodium-glucose co-transporter type 2 (SGLT2) has been proposed as a therapeutic target for type 2 diabetes. However, how DPP-4 inhibitors or SGLT2 inhibitors exert protective actions for diabetic complications in addition to their glucose-lowering effects remains unknown.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetic patients
* Must be able to swallow tablets
* never received DPP-4 inhibitors or SGLT2 inhibitors

Exclusion Criteria:

* uncontrolled diabetes (fasting plasma glucose>200 mg/dL)
* receiving insulin therapy
* hepatic disorders (2.5 fold or greater increases in aspartate transaminase or alanine transaminase levels above the upper limits of normal)
* inflammatory disorders
* neoplastic disorders
* recent (<3months) acute coronary syndrome and stroke
* any acute infection

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Effects of treatment on the nominal change in arterial stiffness from baseline after 6 months of treatment as measured by cardio-ankle vascular index | 6 months of treatment

SECONDARY OUTCOMES:
Change from baseline in subcutaneous and visceral fat volume | 6 months of treatment
Change from baseline in lipid profile including malondialdehyde-modified low-density lipoprotein and remnant-like particle cholesterol | 6 months of treatment
Change from baseline in circulating inflammatory markers | 6 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nobuhiro Tahara, MD, PhD, Study Chair — Department of Medicine, Division of Cardiovascular Medicine, Kurume University School of Medicine
Locations (1):
- Kurume University Hospital, Kurume, Japan

REFERENCES:
- [Derived] Bekki M, Tahara N, Tahara A, Igata S, Honda A, Sugiyama Y, Nakamura T, Sun J, Kumashiro Y, Matsui T, Fukumoto Y, Yamagishi SI. Switching Dipeptidyl Peptidase-4 Inhibitors to Tofogliflozin, a Selective Inhibitor of Sodium-Glucose Cotransporter 2 Improve Arterial Stiffness Evaluated by Cardio-Ankle Vascular Index in Patients with Type 2 Diabetes: A Pilot Study. Curr Vasc Pharmacol. 2019;17(4):411-420. doi: 10.2174/1570161116666180515154555. PMID 29766812